CLINICAL TRIAL: NCT05768412
Title: Radial Artery Access: Demographic Factors Impacting Radial Artery Diameter
Brief Title: Radial Artery Access
Acronym: RADIAL
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Terumo UK Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CFTsp219
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Radiology, Interventional
Keywords: specialty; RADIOGRAPHY, INTERVENTIONAL is available for the diagnostic and therapeutic procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: All patients undergoing Radial Artery Access requiring interventional radiology.
  Interventions: Procedure: Radial Artery Access

INTERVENTIONS:
Procedure: Radial Artery Access — The radial artery is stabilized between the thumb and forefinger of the left hand and 1 to 2 mL of subcutaneous lidocaine is used to create a wheal over the zone of planned entry.

SUMMARY:
This is an imaging investigation to assess the factors effecting radial artery diameter:

* Patient demographics
* Diameter change post standard care preparation

DETAILED DESCRIPTION:
There are significant benefits to radial access intervention, namely superior mortality and morbidity Vs femoral access. In addition, there is significant patient preference and reduced nursing time post procedure in comparison to femoral access supporting day case practice.

Interventional oncology routinely involves repeated procedures therefore patient preference is a key factor in access choice. This again supports day case practice with significant patient preference also noted.

The clinical application of the study is to allow a broader spectrum of procedures to be performed via radial access. Currently due to a limited data available on factors effecting radial artery diameter practice there is a restriction on sheath size use. This limits the procedures that can be performed via this route. By assessing the diameter and factors which increase the vessel, larger access sheaths can be used opening up the procedure portfolio including neuro-interventional procedures and coeliac axis stenting. This will allow these procedures to be performed with added benefits of improved mortality/morbidity in addition patient preference.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or over
2. All patients undergoing Radial Artery Access requiring interventional radiology.

Exclusion Criteria:

1. Prior history of radial artery occlusion
2. Prior history of stroke
3. Need for future dialysis access creation or preservation of upper extremity vasculature for patients with chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients requiring Radial Artery Access at The Christie NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Radial Artery diameter | Before the procedure, during the procedure, and immediately after the procedure
  The change in RA diameter during a standard of care RA access procedure performed by an interventional Radiologist before the procedure, during the procedure and immediately after the procedure and how this compares to patient demographics.

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Najran, Dr, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pending confirmation with funder and PI

REFERENCES:
- [Background] Beyer AT, Ng R, Singh A, Zimmet J, Shunk K, Yeghiazarians Y, Ports TA, Boyle AJ. Topical nitroglycerin and lidocaine to dilate the radial artery prior to transradial cardiac catheterization: a randomized, placebo-controlled, double-blind clinical trial: the PRE-DILATE Study. Int J Cardiol. 2013 Oct 3;168(3):2575-8. doi: 10.1016/j.ijcard.2013.03.048. Epub 2013 Apr 10. PMID 23582415
- [Background] Boyer N, Beyer A, Gupta V, Dehghani H, Hindnavis V, Shunk K, Zimmet J, Yeghiazarians Y, Ports T, Boyle A. The effects of intra-arterial vasodilators on radial artery size and spasm: implications for contemporary use of trans-radial access for coronary angiography and percutaneous coronary intervention. Cardiovasc Revasc Med. 2013 Nov-Dec;14(6):321-4. doi: 10.1016/j.carrev.2013.08.009. Epub 2013 Oct 2. PMID 24095616